CLINICAL TRIAL: NCT05811468
Title: Pilot Study to Evaluate the Correlation Between Peripheral Gene Expression Profile Testing, Tissue-based Gene Expression Profiling, Donor Derived Cell Free DNA, and Histopathology Among High-risk Kidney Transplant Recipients
Brief Title: Study Correlation Between Blood, Tissue Gene Expression, Donor Derived Cell Free DNA and Histopathology in Kidney Transplant Recipients
Status: Withdrawn | Type: Observational
Why Stopped: Trouble enrolling
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Vasil Peev, Physician, Rush University Medical Center
Other Study IDs: 22060707
Record Dates: First submitted 2023-03-17; First posted 2023-04-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Transplant;Failure,Kidney; Kidney Transplant; Kidney Rejection Transplant
Keywords: Gene expression profile; Molecular microscope; Donor derived cell free DNA; Kidney biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will compare the performance of Gene Expression Profile (GEP)/ Donor derived cell free deoxyribonucleic acid (dd-cfDNA) tests, to the following tests: Molecular Microscope (MMDx) and histopathology (study of changes in tissues caused by disease) in their ability to diagnose (exactly identify) various types of injury within the transplanted kidney.

DETAILED DESCRIPTION:
This study will evaluate the performance of the blood-based assays like gene expression panel (GEP), and donor derived cell free DNA (dd-cfDNA) against tissue-based assays like molecular microscope (MMDX) and histopathology in their ability to more accurately detect presence of rejection among kidney transplant recipients deemed at higher than usual risk for immunologic injury i.e., rejection.

Furthermore, the study should shed light on the ability of the different blood- based assays to accurately discern between the different types of rejection (early cellular versus humoral) against such confirmed by histopathology and molecular microscope.

The study will also shed light on the ability of these noninvasive biomarkers to be utilized as a tool of immunomodulation in addition to studying their ability to accurately confirm presence of adequately treated rejection among the recipients of kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a for cause biopsy due to ongoing or suspected "injury" of the allograft.
* Patients will be between 3 months and 7 years post-transplant episode.
* Recipients of both cadaveric and living donor renal transplant are considered eligible.

Exclusion Criteria:

* No multi organ transplant recipients will be included.
* Pregnancy
* HIV positive recipients
* Recipients of kidney transplant from an identical sibling
* Patients with active and biopsy proven BK nephropathy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a for cause biopsy due to ongoing or suspected "injury" of the kidney allograft.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Quantify the number of rejections in the kidney allograft detected via non invasive blood- based testing as reflected in abnormal laboratory readout of GEP value and dd-CFDNA fraction. | Through study completion, an average of 1 year
  The number of rejections in the kidney allograft detected via blood- based non invasive testing will be measured and compared to the number of rejection cases detected by histopathology and MMDX to ascertain accuracy of blood based assays to detect rejection among kidney transplant recipients
Quantify the number of rejection cases detected by histopathology and MMDX as reported by respective pathology laboratories/ pathologists | Through study completion, an average of 1 year
  Measure the number of rejections in the kidney allograft detected by histopathology and MMDX as invasive tests and ascertain concordance of those results with blood based non invasive assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Gupta G, Moinuddin I, Kamal L, King AL, Winstead R, Demehin M, Kang L, Kimball P, Levy M, Bhati C, Massey HD, Kumar D, Halloran PF. Correlation of Donor-derived Cell-free DNA With Histology and Molecular Diagnoses of Kidney Transplant Biopsies. Transplantation. 2022 May 1;106(5):1061-1070. doi: 10.1097/TP.0000000000003838. Epub 2021 May 28. PMID 34075006
- [Background] Park S, Guo K, Heilman RL, Poggio ED, Taber DJ, Marsh CL, Kurian SM, Kleiboeker S, Weems J, Holman J, Zhao L, Sinha R, Brietigam S, Rebello C, Abecassis MM, Friedewald JJ. Combining Blood Gene Expression and Cellfree DNA to Diagnose Subclinical Rejection in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2021 Oct;16(10):1539-1551. doi: 10.2215/CJN.05530421. PMID 34620649
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Sigdel TK, Archila FA, Constantin T, Prins SA, Liberto J, Damm I, Towfighi P, Navarro S, Kirkizlar E, Demko ZP, Ryan A, Sigurjonsson S, Sarwal RD, Hseish SC, Chan-On C, Zimmermann B, Billings PR, Moshkevich S, Sarwal MM. Optimizing Detection of Kidney Transplant Injury by Assessment of Donor-Derived Cell-Free DNA via Massively Multiplex PCR. J Clin Med. 2018 Dec 23;8(1):19. doi: 10.3390/jcm8010019. PMID 30583588